CLINICAL TRIAL: NCT07051980
Title: Feasibility and Safety of Supraglottic Oxygen Delivery Via an Endotracheal Tube for Non-intubated ERCP Anesthesia: A Two-Stage Phase II Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chair of the Department of Anesthesiology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZJU2025B0679
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Choledocholithiasis With Cholecystitis With Obstruction; Obstructive Jaundice; Pancreatitis; Cholelithiasis
Keywords: ERCP; respiratory depression; Hypoxia; Sedation
MeSH Terms: conditions — Jaundice, Obstructive; Pancreatitis; Cholelithiasis; Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supraglottic Oxygen Delivery via an Endotracheal Tube (Experimental): In this group, patients use the Supraglottic Oxygen Delivery via an Endotracheal Tube
  Interventions: Device: Supraglottic Oxygen Delivery via an Endotracheal Tube

INTERVENTIONS:
Device: Supraglottic Oxygen Delivery via an Endotracheal Tube — patients use the Supraglottic Oxygen Delivery via an Endotracheal Tube

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is a technique for evaluating the bile duct, pancreatic duct, and ampulla. Hypoxia is the most common cardiopulmonary complication during ERCP, with a reported rate of 16.2 to 39.2%. The key to preventing hypoxia is to ensure the sufficient oxygenation and ventilation of patients during these procedures. The commonly used approaches to treat hypoxia with a non-instrumented airway are increasing the oxygen flow and lifting the jaw, applying with both hands, displacing the jaw upwards and anteriorly, which allowed the upper airway to remain open. We hypothesized that the supraglottic oxygen delivery via an endotracheal tube can reduce the incidence of hypoxia in patients under deep sedation during ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years；
* The ASA classification ranges from I to III.
* Patients have signed the informed consent form.
* Patients scheduled to undergo sedated ERCP examination;
* The estimated duration of the procedure does not exceed 45 minutes.

Exclusion Criteria:

* Severe cardiac dysfunction (<4 METs);
* Severe renal insufficiency (requiring preoperative dialysis);
* Diagnosed chronic obstructive pulmonary disease (COPD) or other acute/chronic pulmonary diseases requiring long-term/intermittent oxygen therapy;
* Increased intracranial pressure;
* Upper respiratory tract infections (oral/nasal/pharyngeal);
* Fever (core temperature >37.5°C);
* Confirmed pregnancy or current breastfeeding;
* Allergy to sedatives (e.g., propofol) or medical adhesives;
* BMI >30 kg/m²;
* Current participation in other clinical trials;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-12-02 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  75% ≤ SpO2 < 90% for <60 s

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  90% ≤ SpO2 < 95%
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  SpO2 < 75% or 75% ≤ SpO2 < 90% for ≥60 s

OTHER OUTCOMES:
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided